CLINICAL TRIAL: NCT03059290
Title: Incidence of Post-Operative Pain After Single Visit Root Canal Treatment in Necrotic Teeth Using Two Different Rotary Systems (Protaper Nex t& Neolix File)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, karim ahmed abdallah el nahas, master candidate at endodontic department faculty of oral and dental medicine CU, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC-CE-2017-01-15
Record Dates: First submitted 2017-02-12; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Necrotic Pulp
Keywords: post operative pain; Post operative flare ups; Post endodontic pain; Post endodontic flare ups; Necrotic teeth; Non vital teeth; Neolix file; Single rotating file; Protaper next file; Multiple rotating file; Single visit
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- protaper next file (Active Comparator): the PROTAPER NEXT™ X1 (017/04) file, in one or more passes until the working length is reached. Use PROTAPER NEXT X2 (025/06), exactly as described for PROTAPER NEXT X1 file, until the working length is passively reached. Gauge the foramen with a size 025 hand file and, if this file binds at length, the canal is shaped and ready for disinfection. If the size 025 hand file is loose at length, then continue shaping with the PROTAPER NEXT X3 (30/07) and, when necessary, the PROTAPER NEXT X4 (040/06) or PROTAPER NEXT X5 (050/06), gauging after each instrument with the 030, 040 or 050 hand files, respectively. During canal shaping, irrigate, recapitulate with a small-sized hand file after each sequential PROTAPER NEXT instrument, then re-irrigate. in an endodontic motor according to the manufacturer instructions (X-Smart, Dentsply Maillefer, USA.), with torque 2.0 N.cm and speed 300 rpm.
  Interventions: Device: neolix file

INTERVENTIONS:
Device: neolix file — first file used is C1 file size 25 taper 12% as orifice opener and for coronal flaring for 2/3 of canal length the A1 file size 25 taper 8% in narrow or curved canals if size 10 K file (Mani ,Japan ) is loose or pass easily in the canal , but in case of K-file size 20 loose in the canal so we choose large file size 40 taper 4% either of them to the full working length to the full working length with (X-Smart, Dentsply Maillefer, USA.), with speed 300-500 rpm and torque 1.5 N.cm

SUMMARY:
this prospective in vivo randomized clinical is to evaluate the post operative pain (incidence ,degree and duration) with multiple full rotation file (protaper next ®) and single full rotation file (Neolix®) in treating maxillary and mandibular anterior and premolar with chronic pulpitis .Together with our aim from this trial ; we are trying to provide an evidence for the dentists in order to provide the best quality service with the least expenses and thus gaining the patients' trust and saving time, money and effort.

DETAILED DESCRIPTION:
Interventions:

Using neolix file (Ori kam SAS,France)

Control:

Using Protaper next files (Dentsply ,Maillefer , Switzerland)

Treatment in all cases will be completed in one session as follows:

* Full medical and dental history using a schematic dental chart will be obtained from all patients treated during this study. Each tooth will be evaluated for vitality (sensitivity) of pulp tissues using electric pulp tester (Kerr, Analytic Technology Crop, Redmond, WA).
* Patient will be anesthetized; teeth will be isolated with rubber dam.
* Make access and working length will be determined using an electronic apex locator (Root ZX, J.Morita USA, Irvine, CA.) then confirmed with intraoral periapical radiograph, to be 0.5-1 mm, shorter than radiographic apex.
* Cleaning and shaping will be done using crown down preparation technique with rotary files either

  1. neolix file , first file used is C1 file size 25 taper 12% as orifice opener and for coronal flaring for 2/3 of canal length the A1 file size 25 taper 8% in narrow or curved canals if size 10 K file (Mani ,Japan ) is loose or pass easily in the canal , but in case of K-file size 20 loose in the canal so we choose large file size 40 taper 4% either of them to the full working length to the full working length with (X-Smart, Dentsply Maillefer, USA.), with speed 300-500 rpm and torque 1.5 N.cm or
  2. protaper next in sequences by using Prepare straight line access to canal orifice. The ProTaper SX file may be used. Explore the canal using small-sized hand files, determine working length, verify patency and confirm a smooth, reproducible glide path. Always irrigate and if necessary, expand the glide path using small-sized hand files or dedicated mechanical glide path files. Path Files P1 and P2 are recommended. In the presence of NaOCl, brush and follow the glide path, with the PROTAPER NEXT™ X1 (017/04) file, in one or more passes until the working length is reached. Use PROTAPER NEXT X2 (025/06), exactly as described for PROTAPER NEXT X1 file, until the working length is passively reached. Gauge the foramen with a size 025 hand file and, if this file binds at length, the canal is shaped and ready for disinfection. If the size 025 hand file is loose at length, then continue shaping with the PROTAPER NEXT X3 (30/07) and, when necessary, the PROTAPER NEXT X4 (040/06) or PROTAPER NEXT X5 (050/06), gauging after each instrument with the 030, 040 or 050 hand files, respectively. During canal shaping, irrigate, recapitulate with a small-sized hand file after each sequential PROTAPER NEXT instrument, then re-irrigate. in an endodontic motor according to the manufacturer instructions (X-Smart, Dentsply Maillefer, USA.), with torque 2.0 N.cm and speed 300 rpm.
* The rotary files will be introduced inside the canal using EDTA gel "MD-Chelcream, META BIOMED CO.,LTD, Korea".
* The canals will be thoroughly irrigated using 3 ml of 2.5% Sodium hypochlorite between every subsequent instrument. After instrumentation of the canals, paper points will be used for drying.
* Obturation will be carried out using gutta percha cones (25/0.6 or 40/0.4) Or Protaper next cones according to instrument used and canal size with resin sealer (ADSEAL, META BIOMED CO., LTD,Korea).After obturation a cotton pellet will be placed in the pulp chamber and the access cavity will be closed with a temporary filling to avoid coronal leakage. ((MD-Temp, META BIOMED CO., LTD, Korea).
* The patient is given a Numerical Rating Scale and asked to rate his pain level at 6, 12, 24 & 48 hours after obturation.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Patient's age (20-65) years old.
* Upper &lower anterior and premolar teeth diagnosed clinically as necrotic teeth.
* Positive patient's acceptance for participation in the study.
* Sex includes both male and female.
* Patients who can understand Numerical Rating Scale.
* Patients able to sign informed consent.

Exclusion Criteria:

* • Pregnancy or lactation.

  * Medically compromised patients.
  * Patient with multiple teeth that required treatment to eliminate the possibility of pain referral.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
the Incidence of postoperative pain in root canal treatment with necrotic tooth after obturation | 6 hours
the Incidence of postoperative pain in root canal treatment with necrotic tooth after obturation | 12 hours
the Incidence of postoperative pain in root canal treatment with necrotic tooth after obturation | 24 hours
the Incidence of postoperative pain in root canal treatment with necrotic tooth after obturation | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: nehal nabil, assistant professor, Study Chair — faculty of oral and dental medicine - cairo university